CLINICAL TRIAL: NCT03288090
Title: Fatigue After Stroke
Brief Title: Evaluate the Frequency of Fatigue After Cerebral Infarction
Acronym: Fatigue AVC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: Béjot 2017
Record Dates: First submitted 2017-09-18; First posted 2017-09-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Symptomatic Cerebral Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treated
  Interventions: Other: FSS: Fatigue Severity Scale; Other: Neuropsychological evaluation battery; Other: Other functional scores
- Non-treated
  Interventions: Other: FSS: Fatigue Severity Scale; Other: Neuropsychological evaluation battery; Other: Other functional scores

INTERVENTIONS:
Other: FSS: Fatigue Severity Scale — Fatigue scale with 9 items rated from 1 to 7, assessing physical fatigue, fatigue in the psychosocial environment and fatigue in general (3 items in each category).
Other: Neuropsychological evaluation battery — A standardized French neuropsychological battery for the cognitive evaluation of stroke patients.
Other: Other functional scores — Rankin Score, Instrumental Activities of Daily Living (IADL) Score, Rivermead Mobility Index (RMI) scale, Hospital Anxiety Depression scale (HAD) scale for depression / anxiety, Stroke Specific Quality of Life scale for quality of life, Quality Index of Pittsburgh Sleep (PSQI), Vertical Analog Visual Scale for Pain and Vertical Digital Visual Scale

SUMMARY:
Cerebral infarction is a type of stroke that can lead to sometimes disabling sequelae. Among these sequelae, fatigue is frequently reported by patients. It is therefore important for doctors to understand why patients suffer from fatigue after cerebral infarction and to determine whether treatments given for the cerebral infarction may have an impact on this fatigue.

The aim of this research was to study the frequency of fatigue after cerebral infarction, the associated factors, in particular the impact of treatments administered in the acute phase.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting recent symptomatic cerebral infarction (< 1 week) defined according to World Health Organization (WHO) criteria and hospitalised at the Stroke Unit in Dijon University.
* Patients aged 18 years or older.
* Patients who have been informed about the study, or their person of trust for patients unable to express their consent.

Exclusion Criteria:

* Patients (or their person of trust) who refuse to participate in the study.
* Subjects in custody.
* Patients presenting prior co-morbidity as a cause of significant fatigue in the opinion of the investigator
* Patients with dementia or aphasia before the stroke
* Patients (or their person of trust) who may be difficult to contact by telephone during the follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cerebral infarction dating back one week at most
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2018-11-22 (Actual); Study Completion 2018-11-22 (Actual)

PRIMARY OUTCOMES:
Fatigue evaluated using the Fatigue Severity Scale (FSS) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Graber M, Garnier L, Duloquin G, Mohr S, Guillemin S, Ramaget O, Piver A, Tainturier C, Bret-Legrand C, Delpont B, Blanc-Labarre C, Gueniat J, Hervieu-Begue M, Osseby GV, Giroud M, Bejot Y. Association Between Fatigue and Cognitive Impairment at 6 Months in Patients With Ischemic Stroke Treated With Acute Revascularization Therapy. Front Neurol. 2019 Aug 28;10:931. doi: 10.3389/fneur.2019.00931. eCollection 2019. PMID 31555198